CLINICAL TRIAL: NCT00679913
Title: Randomized Controlled Study: Comparison Between Extended and Standard Pancreatoduodenectomy
Brief Title: Standardization of Surgery on the Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sun-Whe Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-0509-513-157
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Pancreaticoduodenectomy; Extended lymphadenectomy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): standard pancreatoduodenectomy
  Interventions: Procedure: Standard pancreatoduodenectomy
- 2 (Active Comparator): extended pancreatoduodenectomy
  Interventions: Procedure: Extended pancreatoduodenectomy

INTERVENTIONS:
Procedure: Standard pancreatoduodenectomy — Standard pancreatoduodenectomy
  Arms: 1
Procedure: Extended pancreatoduodenectomy — Extended pancreatoduodenectomy
  Other Names: Extended lymphadenectomy
  Arms: 2

SUMMARY:
This study was designed to test the hypothesis that more extensive nodal and soft-tissue clearance in patients with adenocarcinoma of the head of the pancreas would improve survival without an increase in morbidity and mortality.

DETAILED DESCRIPTION:
In Japan and in some western treatment centers, there has been a general belief that more extensive surgery may improve outcome for patients with localized, operable pancreatic adenocarcinoma. Initial retrospective reports from centers in Japan suggested that 5-year overall survival rates in patients treated with pancreaticoduodenectomy plus extended lymphadenectomy were higher than those in patients treated by pancreaticoduodenectomy with standard lymphadenectomy. Subsequent prospective randomized trials performed in Europe and the United States failed to confirm a survival benefit from extended lymphadenectomy. Although they failed to confirm a survival benefit from extended lymphadenectomy, the studies had a few pitfalls. The need for Well-designed randomised controlled study is the starting point of our study. This study was designed to test the hypothesis that more extensive nodal and soft-tissue clearance in patients with adenocarcinoma of the head of the pancreas would improve survival without an increase in morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age : 20- 85 years old
* No evidence of metastasis and to be possible to resect radically
* No history of previous radiation therapy or chemotherapy
* Pathological diagnosis: adenocarcinoma of pancreas
* Patients who agree and sign the informed consent
* More than 70 in Karnofsky performance scale

Exclusion Criteria:

* Past medical history of treatment for other malignant disease
* Recurred pancreatic cancer patients
* Patients with R1/R2 resection
* Patients who underwent neoadjuvant chemotherapy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2005-11; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun-Whe Kim, MD., PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Pedrazzoli S, DiCarlo V, Dionigi R, Mosca F, Pederzoli P, Pasquali C, Kloppel G, Dhaene K, Michelassi F. Standard versus extended lymphadenectomy associated with pancreatoduodenectomy in the surgical treatment of adenocarcinoma of the head of the pancreas: a multicenter, prospective, randomized study. Lymphadenectomy Study Group. Ann Surg. 1998 Oct;228(4):508-17. doi: 10.1097/00000658-199810000-00007. PMID 9790340
- [Background] Yeo CJ, Cameron JL, Sohn TA, Coleman J, Sauter PK, Hruban RH, Pitt HA, Lillemoe KD. Pancreaticoduodenectomy with or without extended retroperitoneal lymphadenectomy for periampullary adenocarcinoma: comparison of morbidity and mortality and short-term outcome. Ann Surg. 1999 May;229(5):613-22; discussion 622-4. doi: 10.1097/00000658-199905000-00003. PMID 10235519
- [Background] Farnell MB, Pearson RK, Sarr MG, DiMagno EP, Burgart LJ, Dahl TR, Foster N, Sargent DJ; Pancreas Cancer Working Group. A prospective randomized trial comparing standard pancreatoduodenectomy with pancreatoduodenectomy with extended lymphadenectomy in resectable pancreatic head adenocarcinoma. Surgery. 2005 Oct;138(4):618-28; discussion 628-30. doi: 10.1016/j.surg.2005.06.044. PMID 16269290
- [Background] Michalski CW, Kleeff J, Wente MN, Diener MK, Buchler MW, Friess H. Systematic review and meta-analysis of standard and extended lymphadenectomy in pancreaticoduodenectomy for pancreatic cancer. Br J Surg. 2007 Mar;94(3):265-73. doi: 10.1002/bjs.5716. PMID 17318801
- [Derived] Jang JY, Kang MJ, Heo JS, Choi SH, Choi DW, Park SJ, Han SS, Yoon DS, Yu HC, Kang KJ, Kim SG, Kim SW. A prospective randomized controlled study comparing outcomes of standard resection and extended resection, including dissection of the nerve plexus and various lymph nodes, in patients with pancreatic head cancer. Ann Surg. 2014 Apr;259(4):656-64. doi: 10.1097/SLA.0000000000000384. PMID 24368638

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2006 and November 2009, 244 patients were enrolled in this study, after excluding the 9 patients who refused to participate after initial agreement. After enrollment, 44 patients were excluded due to having unresectable or metastatic tumors, as determined intraoperatively
Pre-assignment Details: After enrollment, some patients were excluded due to (1) unresectable condition or metastasis found during surgery; (2) surgical rule violation; (3) inadequate case report form; or (4) pathologic diagnosis other than conventional ductal adenocarcinoma.
Groups:
- Standard Pancreatoduodenectomy: standard pancreatoduodenectomy Standard pancreatoduodenectomy: Standard pancreatoduodenectomy In standard resection, the lymph nodes around the pancreas head (LN 13, 17) and gallbladder (LN 12c) were removed without nerve dissection around the hepatic or superior mesenteric artery (SMA)
- Extended Pancreatoduodenectomy: extended pancreatoduodenectomy Extended pancreatoduodenectomy: Extended pancreatoduodenectomy During extended resection, the lymph nodes around the common hepatic artery (LN 8), celiac axis (CA) (LN 9), peripancreatic area (LN 13, 17), hepatoduodenal ligament (LN 12), SMA (LN 14) and paraaortic area (LN16) between the CA and inferior mesenteric artery were dissected. All soft tissues around the hepatoduodenal ligament were completely dissected and skeletonized. The nerve plexus or ganglion on the right side of the CA and SMA was dissected semi-circumferentially.
Period: Overall Study
Arm/Group | Standard Pancreatoduodenectomy | Extended Pancreatoduodenectomy
Started | 101 | 99
Completed | 83 | 86
Not Completed | 18 | 13
Not completed — Protocol Violation | 18 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Pancreatoduodenectomy | Extended Pancreatoduodenectomy | Total
Number analyzed (Participants) | 83 | 86 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8.7) | 63.4 (9.5) | 62.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 42 | 76
  Male | 49 | 44 | 93

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: comparison of 2-year overall survival rate between standard and extended pancreaticoduodenectomy; number of surviving participants 2 years after surgery
Time Frame: 2 year after surgery
Measure: Number; unit: participants
Arm/Group | Standard Pancreatoduodenectomy | Extended Pancreatoduodenectomy
Number analyzed (Participants) | 83 | 86
participants | 37 | 31

2. Secondary Outcome: Morbidity
Description: Number of participants with morbidity, such as bleeding, sepsis, pancreatic fistula, intra-abdominal abscess, wound infection, delayed gastric emptying, and diarrhea after standard and extended pancreaticoduodenectomy
Time Frame: within 2 years after surgery
Measure: Number; unit: participants
Groups:
- Extended Pancreatoduodenectomy: extended pancreatoduodenectomy
  Extended pancreatoduodenectomy: Extended pancreatoduodenectomy During extended resection, the lymph nodes around the common hepatic artery (LN 8), celiac axis (CA) (LN 9), peripancreatic area (LN 13, 17), hepatoduodenal ligament (LN 12), SMA (LN 14) and paraaortic area (LN16) between the CA and inferior mesenteric artery were dissected. All soft tissues around the hepatoduodenal ligament were completely dissected and skeletonized
Arm/Group | Standard Pancreatoduodenectomy | Extended Pancreatoduodenectomy
Number analyzed (Participants) | 83 | 86
participants | 27 | 37

ADVERSE EVENTS:
Time Frame: every 3 months after surgery
Arm/Group | Standard Pancreatoduodenectomy | Extended Pancreatoduodenectomy
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/86
Other Adverse Events (participants affected / at risk) | 0/83 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: embargo of 60 days or less